CLINICAL TRIAL: NCT00352235
Title: Phase I/II Trial of KRN7000 in Patients With Chronic Hepatitis C Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: KRN7000 HCV
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2006-07-14 (Estimated); Status verified 2006-07

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; KRN7000; a-GalCer; immunotherapy; Natural Killer T cells; interferon
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — KRN 7000

INTERVENTIONS:
Drug: KRN7000

SUMMARY:
Phase I/II trial of KRN7000 in patients with chronic hepatitis C.

Study objectives: To evaluate and compare the safety and tolerability of 3 ascending doses of a-GalCer.

The primary efficacy parameter: HCV-RNA response at the end of treatment. Secondary efficacy parameter: Serum ALT response. Further objectives of the study are to evaluate the effect of a-GalCer on serum cytokines IFNg and TNFa and on iNKT cells.

Number of dose levels: 3 Investigational product: KRN7000 Route of administration: intravenous Dosages and frequency: 0.1, 1, 10 mcg/kg, monthly injection, 3 times (day 0, day 28 and day 56)

DETAILED DESCRIPTION:
Phase I/II trial of KRN7000 in patients with chronic hepatitis C.

This study is a multicenter double-blind randomized placebo-controlled phase I/II dose-escalation trial. The protocol is conducted in The Netherlands, Belgium and Germany. Patients with chronic hepatitis C who met the inclusion criteria are assigned to receive a-GalCer (KRN7000 ((2S, 3S, 4R)-1-O-(a-D-galactopyranosyl)-N-hexacosanoyl-2-amino-1,3,4-octadecanetriol), Kirin Pharmaceutical Co., Ltd., Gunma, Japan) or placebo intravenously, thrice with intervals of 4 weeks. Cohorts of 12 patients are entered at each of the three dose levels (0.1, 1 and 10 mg/kg body weight). Three patients per dose level are randomized to the placebo arm.

Dose escalation to the next cohort are decided after evaluation by a safety review board of all the safety data collected on all the patients who had completed 3 weeks after the first injection in the preceding dose cohort. After completion of 8 weeks of treatment, with injections at 0, 4 and 8 weeks, patients are monitored without further therapy for an additional 16 weeks.

Study objectives: The objective of the study is to evaluate and compare the safety and tolerability of 3 ascending doses of a-GalCer. The primary efficacy parameter is the response at the end of treatment, based on serum hepatitis C virus ribonucleic acid (HCV RNA) levels. As a secondary efficacy parameter serum ALT levels are evaluated. Further objectives of the study are to evaluate the effect of a-GalCer on serum cytokines IFNg and TNFa and on iNKT cells.

ELIGIBILITY:
Inclusion Criteria:

Chronic hepatitis C Liver biopsy within 3 years of entry into the study HCV RNA > 10000 copies/mL Age 18-70 years ALT > 1.2 times ULN written informed consent Adequate contraception

Exclusion Criteria:

Cirrhosis Decompensated liver disease ALT > 10 times ULN Pregnancy Major other illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2003-08; Study Completion 2005-05

PRIMARY OUTCOMES:
Decrease in serum hepatitis C virus ribonucleic acid (HCV RNA) levels.

SECONDARY OUTCOMES:
Normalization of serum ALT levels.
Effect on serum cytokines IFNg and TNFa and on iNKT cells.

CONTACTS AND LOCATIONS:
Overall Officials: Carin MJ van Nieuwkerk, MD, PhD, Principal Investigator — VU medical Center, Amsterdam
Locations (1):
- Erasmus MC, Rotterdam, Netherlands